CLINICAL TRIAL: NCT03982173
Title: A Phase II Whole Exome Sequencing-based Basket Trial for Combination Therapy With Durvalumab (Anti-PDL1) (MEDI4736) and Tremelimumab (Anti-CTLA4) in Patients With Metastatic Solid Tumors
Brief Title: Basket Trial for Combination Therapy With Durvalumab (Anti-PDL1) (MEDI4736) and Tremelimumab (Anti-CTLA4) in Patients With Metastatic Solid Tumors
Acronym: MATILDA
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Similar clinical trials showed not very encouraging results, which made us decide, after several modifications to the protocol and numerous difficulties encountered, to abandon the trial.
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018-003115-21; 2018/2798 (Other: CSET number)
Record Dates: First submitted 2019-06-07; First posted 2019-06-11 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Metastatic Colorectal Cancer; Triple Negative Breast Cancer; Prostate Adenocarcinoma; Stomach Adenocarcinoma; Esophageal Adenocarcinoma
MeSH Terms: conditions — Colorectal Neoplasms; Triple Negative Breast Neoplasms; Adenocarcinoma Of Esophagus | interventions — tremelimumab; durvalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- previously treated patients with solid tumors (Experimental): previously treated patients with solid tumors harboring a high mutational load.
  Interventions: Drug: Tremelimumab; Drug: Durvalumab

INTERVENTIONS:
Drug: Tremelimumab — tremelimumab 75mg
Drug: Durvalumab — Durvalumab 1500mg

SUMMARY:
To determine the efficacy (as measured by overall tumour response rate) of the combination of durvalumab and tremelimumab when given to previously treated patients with solid tumors harboring a high mutational load.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent obtained from the subject prior to performing any protocol-related procedures, including screening evaluations
2. Age ≥ 18 years
3. Histologically confirmed diagnosis of metastatic colorectal adenocarcinoma (without microsatellite instability (not MSI), triple negative breast cancer, prostate adenocarcinoma and stomach and esophageal gastric junction adenocarcinoma.
4. Metastatic disease or unresectable locally advanced malignancy that is resistant or refractory to standard therapy or for which standard therapy does not exist or is not considered appropriate by the Investigator
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 with no deterioration over the 2 weeks prior to starting dose
6. Estimated life expectancy of greater than 12 weeks
7. Detection of ≥ 5 somatic mutations per megabase measured by whole exome sequencing in a tumor sample of the patient taken after completing last therapy, within a molecular screening program (this data must been known before screening period)
8. Total bilirubin ≤ 1.5 ULN (for subjects with documented/suspected Gilbert's disease, bilirubin ≤ 3 ×ULN), ALT or AST ≤ 2.5 ULN (for subjects with liver metastases, AST or ALT ≤ 5 × ULN), albumin ≥ 30 g/L
9. Haemoglobin > 9 g/dL, neutrophils > 1500/mm3, platelets > 100,000/mm3
10. Serum creatinine CL>40 mL/min by the Cockcroft-Gault formula (Cockcroft and Gault 1976) or by 24-hour urine collection for determination of creatinine clearance.
11. At least one lesion, not previously irradiated, which can be measured at baseline as ≥10 mm in the longest diameter (except lymph nodes which must have short axis ≥ 15 mm) with computed tomography (CT) or magnetic resonance imaging (MRI) and suitable for repeated assessment according to Response Evaluation Criteria in Solid Tumors (RECIST) guidelines v1.1.
12. Females of childbearing potential who are sexually active with a non-sterilized male partner must use at least 1 highly effective method of contraception, from screening, and must agree to continue using such precautions for 180 days after the final dose of durvalumab and tremelimumab or 90 days after the last dose of durvalumab monotherapy, whichever is the longer time period; cessation of birth control after this point should be discussed with a responsible physician. Male partners of a female subject must use male condom plus spermicide throughout this period. Not engaging in sexual activity for the total duration of the drug treatment and the drug washout period is an acceptable practice; however, periodic abstinence, the rhythm method, and the withdrawal method are not acceptable methods of birth control.

    1. Females of childbearing potential are defined as those who are not surgically sterile (ie, bilateral tubal ligation, bilateral oophorectomy, or complete hysterectomy) or postmenopausal (defined as 12 months with no menses without an alternative medical cause)
    2. Subjects must use at least one method of contraception highly effective, such as Copper T intrauterine device, Levonorgestrel-releasing intrauterine system (eg, Mirena® ) a Etonogestrel implants; eg, Implanon or Norplan, Intravaginal device; eg, ethinylestradiol and etonogestrel, Medroxyprogesterone injection: DepoProvera, Normal and low dose combined oral contraceptive pil, Norelgestromin/ethinylestradiol transdermal system or use of Cerazette (desogestrel)
    3. Female subjects should also refrain from breastfeeding throughout this period
    4. Females of childbearing potential must have a negative serum pregnancy test result within 3 days prior to initiation of study drugs Nonsterilized males who are sexually active with a female partner of childbearing potential must use a male condom with spermicide for 180 days after the final dose of durvalumab and tremelimumab or 90 days after the last dose of durvalumab monotherapy, whichever is the longer time period. Female partners of a male subject must use a highly effective method of contraception throughout this period. Not engaging in sexual activity is an acceptable practice; however, occasional abstinence, the rhythm method, and the withdrawal method are not acceptable methods of contraception. Male subjects should refrain from sperm donation and female subjects should refrain from oocyte donation throughout this period.
13. Absence of any psychological, familial or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before inclusion in the trial
14. Patient must be affiliated to a social security system or beneficiary of the same

Exclusion Criteria:

1. Participation in another clinical study with an investigational product during the last 4 weeks (excepting noninterventional clinical studies)
2. Concurrent enrolment in another clinical study (with an investigational product), unless it is an non-interventional clinical study
3. Any previous treatment with immunotherapy including (but not limited to) compounds such as, PD1 or PD-L1 inhibitors, including durvalumab or an anti-CTLA4 inhibitors, including tremelimumab.
4. Previous exposure to anti oncogenic vaccines, such as Sipuleucel - T is not allowed
5. History of another primary malignancy except for:

   1. Malignancy treated with curative intent and with no known active disease ≥5 years before the first dose of study drug and of low potential risk for recurrence
   2. Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
   3. Adequately treated carcinoma in situ without evidence of disease eg, cervical cancer in situ.
6. Receipt of the last dose of anti-cancer therapy (chemotherapy, endocrine therapy, targeted therapy, biologic therapy, tumor embolization, monoclonal antibodies, other investigational agent) 28 days prior to the first dose of study drug. A shorter duration of five half times may be considered after Sponsor approval, for patients treated with non-cytotoxic drugs). (If sufficient wash-out time has not occurred due to the schedule or PK properties of an agent, a longer wash-out period may be required.)
7. Current or prior use of immunosuppressive medication within 14 days before the first dose of durvalumab or tremelimumab. The following are exceptions to this criterion:

   1. Intranasal, inhaled, topical steroids, or local steroid injections (eg, intra articular injection)
   2. Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or its equivalent
   3. Steroids as premedication for hypersensitivity reactions (eg, CT scan premedication)
8. Any unresolved toxicity NCI CTCAE Grade ≥2 from previous anticancer therapy with the exception of alopecia, vitiligo, and the laboratory values defined in the inclusion criteria

   1. Patients with Grade ≥2 neuropathy will be evaluated on a case-by-case basis after consultation with the Study Physician.
   2. Patients with irreversible toxicity not reasonably expected to be exacerbated by treatment with durvalumab or tremelimumab may be included only after consultation with the Study Physician.
9. Any concurrent chemotherapy, IMP, biologic, or hormonal therapy for cancer treatment. Concurrent use of hormonal therapy for non-cancer-related conditions (eg, hormone replacement therapy) is acceptable.
10. Major surgical procedure (as defined by the Investigator) within 28 days prior to the first dose of IMP. Note: Local surgery of isolated lesions for palliative intent is acceptable.
11. Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [eg, colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc]). The following are exceptions to this criterion:

    1. Patients with vitiligo or alopecia
    2. Patients with hypothyroidism (eg, following Hashimoto syndrome) stable on hormone replacement
    3. Any chronic skin condition that does not require systemic therapy
    4. Patients without active disease in the last 5 years may be included but only after consultation with the study physician
    5. Patients with celiac disease controlled by diet alone
12. History of primary immunodeficiency
13. History of allogeneic organ transplant
14. Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the patient to give written informed consent
15. Past medical history of ILD, drug-induced ILD, radiation pneumonitis which required steroid treatment, or any evidence of clinically active interstitial lung disease
16. Active infection including tuberculosis (clinical evaluation including clinical history, physical examination and radiographic findings, and TB testing in line with local practice), hepatitis B (known positive HBV surface antigen (HBsAg) result), hepatitis C, or human immunodeficiency virus (positive HIV 1/2 antibodies). Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. Patients positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
17. History of leptomeningeal carcinomatosis
18. Subjects with uncontrolled seizures
19. Brain metastases or spinal cord compression unless the patient is stable (asymptomatic; no evidence of new or emerging brain metastases; and stable and off steroids for at least 28 days prior to start of study treatment). Following radiotherapy and/or surgery of the brain metastases patients must wait 4 weeks following the intervention and before randomisation with imaging to confirm stability.
20. Receipt of live attenuated vaccine within 30 days prior to the first dose of IMPs. Note: Patients, if enrolled, should not receive live vaccine whilst receiving IMPs and up to 30 days after the last dose of IMPs.
21. Female patients who are pregnant or breastfeeding or male or female patients of reproductive potential who are not willing to employ effective birth control from screening to 180 days after the last dose of durvalumab + tremelimumab combination therapy or 90 days after the last dose of durvalumab monotherapy or confirmation of PD and investigator determination that the subject is no longer benefiting from treatment with durvalumab + tremelimumab whichever is the longer time period.
22. Known allergy or hypersensitivity to any of the study drugs or any of the study drug excipients.
23. Any condition that, in the opinion of the investigator, would interfere with evaluation of study treatment or interpretation of patient safety or study results
24. Patient under guardianship or deprived of his liberty by a judicial or administrative decision or incapable of giving its consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-09 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2024-12-05 (Estimated)

PRIMARY OUTCOMES:
Objective tumour response rate | at 12 weeks
  measured according to RECIST (version 1.1)

IPD SHARING:
Plan to Share IPD: Undecided